CLINICAL TRIAL: NCT05209087
Title: Effects of Parental Influence on Physical Activity Level And Participation in Children With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Serenay Zorlu, Graduate Student, Hacettepe University
Other Study IDs: 16969557-451
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: duchenne muscular dystrophy; physical activity participation; parental influence; physical activity level
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Duchenne Muscular Dystrophy: Children with Duchenne Muscular Dystrophy who are between Levels 1-4 (continuing ambulation) according to Brooke Lower Extremity Functional Classification will be included in the study. This classification method was designed on the basis of the classification method to determine the functional status of the lower and upper extremities in the clinical evaluation of Duchenne Muscular Dystrophy.

SUMMARY:
This study was planned to investigate the parental influence on physical activity (PA) level and participation in ambulatory children with Duchenne muscular dystrophy (DMD). For this purpose, 30 children with DMD between the ages of 8-18, who were between Levels 1-4 according to the Brooke Lower Extremity Functional Classification (BLEFC), were included in the study. The demographic information of the participants and their detailed information about the disease were recorded. Parents' PA level was assessed via International Physical Activity Questionnaire-Short Form (IPAQ-SF); Children's PA level was assessed via Physical Activity Questionnaire for Children (PAQ-C) and pedometer, participation was assessed via Pediatric Outcomes Data Collection Instrument (PODCI), and parental influence was assessed via Children's Physical Activity Correlates (CPAC). Additionally, children's PA interest was assessed via Children's Attraction to Physical Activity (CAPA). SPSS 25 program was used in the statistical analysis of the evaluation results. The mean age of the individuals included in the study was found to be 8,70±0,84. Parental influence evaluations, positive and weak-moderate correlations were determined between CPAC Questionnaire "Parental Influence" sub-dimension with PAQ-C (r=0,582), CAPA (0,432) and PODCI (r=0,372) (p<0,05). A positive, moderate correlation was found between the PA levels of mothers obtained from IPAQ-SF and PAQ-C (p<0,01). The results of the study show that the parents, especially the mother who is the primary caregiver, can be an important factor to improve the PA levels, increase their attraction to PA and participation in children with DMD.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is the most common neuromuscular disease in childhood with an incidence of 1 per 3600-6000 live male births worldwide. It shows X-linked recessive inheritance. It is caused by a mutation in the gene encoding the dystrophin protein localized in Xp21.2. It is characterized by complete or partial deficiency of the cell membrane protein called dystrophin. Deficiency of dystrophin causes disruption of the structure of the muscle sarcolemma. Accordingly, the stress caused by repetitive contractions damages the sarcolemma. This deficiency leads to continuous degeneration of muscle fibers. As a result, it causes progressive loss in the strength of skeletal muscles, respiration and later cardiac muscles. As the disease progresses, due to muscle damage and weakness, the child's ability to perform daily tasks such as climbing stairs and walking short distances becomes impaired and functional skills decrease. Respiratory and cardiac muscle involvement is the most important cause of mortality in these patients before the age of 30.

Participation is a measurable outcome of health. This measure is defined as direct participation in life by the International Classification of Functioning, Disability and Health (ICF). Participation for children and youth includes activities such as personal care, mobility, social relations, education, play and leisure activities. Disabled children participate less in daily activities than healthy children.

Considering the progression of their diseases, the participation of children with DMD in physical activity decreases over time. Functional disorders in children with DMD affect their daily living activities, limiting their participation in similar activities with their peers. Research shows that children with DMD have lower levels of physical activity from a young age than their healthy peers. There are also studies in the literature showing that there is a decrease in the functional independence and quality of life of children with DMD as well as their families and caregivers.

Participation in regular physical activity in disabled children and youth contributes to physical, psychosocial and social development. Safe and effective physical activity can positively affect the nutritional status, mobility and social participation of patients with DMD throughout their lives. This indicates that we need to improve our understanding of the determinants and mechanisms underlying the thinking of children and adolescents with DMD regarding physical activity behaviors.

Parents play an important role in shaping their children's beliefs, attitudes, and behaviors across a wide range of developmental domains, including cognitive, social, and emotional domains. In addition to studies examining physical activity interventions for healthy children and youth, strong evidence has been shown that families can have a significant influence in increasing the physical activity of children and youth with disabilities. Parental behaviors that promote physical activity in children have two aspects: 1) role modeling, which includes efforts to be active alongside the parent's interest in physical activity, and 2) parental encouragement and involvement, providing access and opportunities for the child to be active (for example transport to sports complexes and parks). Studies examining the influence of parents on physical activity behaviors of children and adolescents shows that there is a positive relationship between parental behaviors and the activities in which children participate.

When the literature on individuals with DMD was examined, a limited number of studies were found that investigated both the physical activity level of the child with DMD and the effects of the parent on the activity level of the child with DMD. Therefore, the aims of our study are to determine the physical activity levels of school-age children with Duchenne Muscular Dystrophy who can walk and to investigate the effect of the family on the child's physical activity level and participation.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the study on a voluntary basis
* The ages of 8 and 18 who have been diagnosed with Duchenne Muscular Dystrophy
* Being in the first four levels according to the Brooke Lower Extremity Functional -Classification (BAEFS) (ambulatory children)
* Not having difficulties in cooperation

Exclusion Criteria:

* Have undergone any musculoskeletal surgery in the last 6 months that may affect gait
* Having compliance problems that cannot follow the physiotherapist's instructions

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hacettepe University Faculty of Physical Therapy and Rehabilitation Pediatric Neuromuscular Diseases Unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire-Short Form-IPAQ-SF | Baseline
  The International Physical Activity Questionnaire-Short Form is used to determine the physical activity level of parents between the ages of 18-65. It contains 7 questions about the activities done in the last 7 days.
Physical Activity Questionnaire for Children-PAQ-C | Baseline
  The Physical Activity Questionnaire for Children is used to determine the physical activity level of children between the ages of 8-14. It contains 7 questions about the activities done in the last 7 days.
Physical Activity Questionnaire for Adolescents-PAQ-A | Baseline
  The Physical Activity Questionnaire for Adolescents is used to determine the physical activity level of children between the ages of 14-18. It contains 7 questions about the activities done in the last 7 days.
Six Minute Walk Test-6MWT | Baseline
  Six Minute Walk Test is used to measure walking function and physical capacity at the submaximal level in children with DMD. 6MWT is used as the gold standard in evaluating the functional capacity of patient with Duchenne Muscular Dystrophy.
North Star Ambulatory Assessment-NSAD | Baseline
  North Star Ambulatory Assessment is a performance-based test developed to evaluate the ambulation level of children with DMD who can walk.
Children's Attraction to Physical Activity Scale-CAPA | Baseline
  Children's Attraction to Physical Activity Scale is a questionnaire that used to assess children's interest in physical activity. It consists of 15 questions. The questionnaire is filled by the researcher reading the questions aloud and the child responding.
The Pediatric Outcomes Data Collection Instrument (PODCI) | Baseline
  The Pediatric Outcomes Data Collection Instrument is a questionnaire used to measure functional outcomes. Functional dimensions assessed include upper extremity functioning, transfers and basic mobility, sports and physical function, comfort/pain, global function and happiness with physical condition. This study uses PODCI to quantify the physical activity participation of a group of DMD patients.
Pedometer | 5 days
  Pedometers are measurement tools developed for counting steps that can measure and record vertical movements. This study used pedometer to determine the physical activity level of children.
Children's Physical Activity Correlates-CPAC | Baseline
  Children's Physical Activity Correlates used to evaluate the factors affecting physical activity in children. It consists of 44 questions. The questionnaire is filled by the researcher reading the questions aloud and the child responding.

CONTACTS AND LOCATIONS:
Overall Officials: İpek Gürbüz, Assoc. Prof., Study Chair — Hacettepe University; Serenay Zorlu, Principal Investigator — Medipol University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)